CLINICAL TRIAL: NCT04779502
Title: The Efficacy of Oregano Essential Oil in Reducing Oral Halitosis :A Randomized Controlled Trial
Brief Title: The Efficacy of Oregano Essential Oil in Reducing Oral Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MOHAMED SAEED M. ALI (Other)
Responsible Party: Sponsor-Investigator, MOHAMED SAEED M. ALI, Principal Investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 131619
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Halitosis
Keywords: oral halitosis; oregano essential oil; mouthwash
MeSH Terms: conditions — Halitosis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- oregano (Experimental): oregawash mouthwash was used twice times daily for 7 days
  Interventions: Other: oregawash
- placebo (Placebo Comparator): distilled water was used twice times daily for 7 days
  Interventions: Other: placebo
- chlorhexidine (Active Comparator): Corsodyl with 0.2%CHX mouthwash was used twice times daily for 7 days
  Interventions: Other: corsodyl

INTERVENTIONS:
Other: oregawash — mouthwash containing oregano essential oil
  Arms: oregano
Other: corsodyl — 0.2% chlorhexidine mouthwash
  Other Names: chlorhexdine
  Arms: chlorhexidine
Other: placebo — distilled water
  Other Names: distilled water
  Arms: placebo

SUMMARY:
the efficacy of commercially available oregano essential oil mouthwash in the reduction of oral halitosis was compared to chlorhexidine and distilled water and the results showed significant reduction of organoleptic tongue and floss scores and BANA test scores compared to placebo

DETAILED DESCRIPTION:
the results showed that oregawash showed a comparable effect to chx in reducing oral halitosis

ELIGIBILITY:
Inclusion Criteria:

1. Organoleptic score was >2 at baseline.
2. Participants between 18-23 years of age.
3. The subjects had no systemic disease and were not taking antibiotics or receiving other antimicrobial therapy.
4. The subjects did not receive the same time treatment for their halitosis.

Exclusion Criteria:

1. Smokers, alcoholics and drug addicts.
2. Patients with periodontitis or pocket depth >6 mm.
3. Patients taking drugs which induced xerostomia.
4. Subjects consuming spicy food: garlic or onions two days before examination.
5. Patients with orthodontic appliances or removable dentures.
6. pregnancy

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
organoleptic tongue and floss scores | 9 month
  organoleptic measuements

SECONDARY OUTCOMES:
BANA test | 9 month
  chair side BANA test

CONTACTS AND LOCATIONS:
Overall Officials: mohamed s albana, director, Principal Investigator — univeristy of baghdad
Locations (1):
- Univeristy of Baghdad, Baghdad, Rasafa, Iraq

IPD SHARING:
Plan to Share IPD: No